CLINICAL TRIAL: NCT07266298
Title: A Phase I, Multicenter, Dose-escalation, Single-arm Study of PRAME Antigen-targeted TCR-T Cells(NW-101C) in the Treatment of Subjects With Advanced Solid Malignant Tumors.
Brief Title: TCR-engineered T Cells (NW-101C) in Patients With Solid Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neowise Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NW-101C-002
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Solid Metastatic Tumor

STUDY DESIGN:
Intervention Model Description: A classic 3+3 model will be used to dose escalation,4 doses will be used: 4×10^8±30%, 8×10^8±30%, 15×10^8±30% and 30×10^8±30% TCR-T cells/ patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NW-101C dose 1-4 (Experimental)
  Interventions: Biological: NW-101C

INTERVENTIONS:
Biological: NW-101C — 4 dosage of NW-101C will be tested in this study using classic 3+3 dose escalation approach: 4×10^8±30%, 8×10^8±30%,15×10^8±30% and 30×10^8±30% TCR-T+ cells

SUMMARY:
This clinical trial is a prospective, dose-escalation, multicenter, single- arm, Phase 1 clinical trial to evaluate the safety, tolerability, PK and preliminary clinical activity of PRAME Antigen-targeted TCR-T Cells (NW-101C) infusion in patients with previously heavily treated, metastatic solid malignant tumors.

DETAILED DESCRIPTION:
Using a classic 3+3 dose escalation design, this study will enroll ~24 subjects to characterize the safety and preliminary anti-tumor activity of NW-101C.

SCREENING: Patient eligibility will be determined by protocol inclusion/exclusion criteria including HLA (human leukocyte antigen) and a biopsy (or collection of archival tumor tissue) for biomarker screening. Leukapheresis for potential manufacturing of the NW-101C cellular product may be performed,if patients are HLA-A*02:01 positive and meet the eligibility criteria for leukapheresis.

MANUFACTURING: NW-101C products will be made from the patients' white blood cells.

TREATMENT: Lymphodepletion with cyclophosphamide and fludarabine will occur in the days before the NW-101C product infusion to improve the duration of time that NW-101C product stays in the body. The patient will be admitted to the hospital during the T-cell infusion until 28 days following NW-101C infusion. After the NW-101C product infusion, dose -limiting toxicities (DLT) will be assessed from the infusion of NW-101C until 28 days following the infusion of NW-101C.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years
* Diagnosis of pathologically or histologically confirmed unresectable or advanced solid tumors and must have no standard treatment options available or unable to tolerate the currently available standard treatments
* For patients with ovarian caner :Patients must have confirmed diagnosis of Platinum-resistant ovarian epithelial carcinoma(PROC)
* HLA-A*02:01positive
* Patient's tumor must express PRAME assessed by central lab,Retrospective testing will be required for patients that qualify.
* Adequate organ function prior to apheresis and lymphodepleting chemotherapy
* ECOG performance status of 0-1
* At least one tumor lesion measurable according to RECIST 1.1

(Additional protocol-defined Inclusion criteria may apply)

Exclusion Criteria:

* Received the following treatments: Cytotoxic chemotherapy within 2 weeks prior to apheresis and within 1 week prior to lymphodepletion; Treatment with antibodies (including but not limited to those with monoclonal antibodies and immune checkpoint inhibitors) or other biologic therapy within 2 weeks prior to apheresis and within 1 week prior to lymphodepletion; Immunosuppressive agents (e.g., calcineurin inhibitors, methotrexate or other chemotherapeutic agents, mycophenolate mofetil, rapamycin, thalidomide, immunosuppressive antibodies such as anti-TNF, anti-IL-6, or anti-IL-6 receptor) within 2 weeks prior to apheresis and within 1 week prior to lymphodepletion
* History of allergic reactions to cyclophosphamide, fludarabine, or any other chemical or biological components of the drugs used in this study
* History of chronic or recurrent severe autoimmune disease, or active immune disease requiring treatment with steroids or other immunosuppressive agents within 1 year prior to enrollment
* Have symptomic CNS metastases
* Have leptomeningeal disease or carcinomatous meningitis
* Have ongoing or active infection
* Active infections with HIV, HBV, HCV, or syphilis
* Breastfeeding or pregnant

(Additional protocol-defined Exclusion criteria may apply)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Dose-limiting toxicities(DLTs) of NW-101C in patients with solid malignant tumors | 28 days following NW-101C infusion
  Type, frequency and severity of adverse events assessed by CTCAE5.0
Evaluate the Maximum Tolerated Dose (MTD) of NW-101C in patients with solid malignant tumors | Through the study completion, an average of 2 years
  Type, frequency and severity of adverse events assessed by CTCAE5.0

SECONDARY OUTCOMES:
Evaluate the AUC of NW-101C in patients with solid malignant tumors | 2 years following NW-101C infusion
  Area under the Plasma concentration versus time curve(AUC) assessed centrally
Evaluate the Objective response rate (ORR) of NW-101C in patients with solid malignant tumors | 2 years following NW-101C infusion
  Complete response (CR) and partial response (PR) assessed by investigators following RECIST1.1 criteria
Evaluate the Cmax of NW-101C in patients with solid malignant tumors | Through the study completion, an average of 2 years
  Maximum Concentration(Cmax) assessed centrally
Evaluate the Tmax of NW-101C in patients with solid malignant tumors | Through the study completion, an average of 2 years
  Time of Maximum Concentration assessed centrally

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No